CLINICAL TRIAL: NCT05377606
Title: Macular Perfusion and Sensitivity Following Silicone Oil Tamponade Versus SF6 Gas for Primary Rhegmatogenous Retinal Detachment
Brief Title: Primary Vitrectomy With Silicone Oil or SF6 for Rhegmatogenous Retinal Detachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Safe Abdelmesih Abdelmalak, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-187-2021
Record Dates: First submitted 2022-02-13; First posted 2022-05-17 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Rhegmatogenous Retinal Detachment; Primary Vitrectomy
MeSH Terms: interventions — Silicone Oils

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Surgeon will be masked to the tamponading agent (silicone oil or gas) till the end of the operation when either agent will be injected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silicone oil group (Active Comparator): Primary pars plana vitrectomy will be performed and silicone oil will be used as the tamponading agent. For these patients, optical coherence tomography (OCT) and angiography (OCTA), along with microperimetry will be done 2 months after the primary surgery. Then they will be scheduled for silicone oil removal after 3 months from the time of primary surgery. Finally, the OCT, OCTA, and microperimetry will be repeated once more after 4 months from the vitrectomy (i.e. one month after the silicone oil removal).
  Interventions: Procedure: Pars plana vitrectomy with silicone oil
- Sulfur hexafluoride (SF6) group (Active Comparator): Primary pars plana vitrectomy will be performed and sulfur hexafluoride (SF6) will be used as the tamponading agent. For these patients, optical coherence tomography (OCT) and angiography (OCTA), along with microperimetry will be done 2 months and 4 months after the primary surgery.
  Interventions: Procedure: Pars plana vitrectomy with SF6

INTERVENTIONS:
Procedure: Pars plana vitrectomy with silicone oil — Silicone oil will be used at the end of primary vitrectomy. OCT, OCTA and microperimetry will be done 2 months later. Silicone oil will be removed at 3 months. Finally, the OCT, OCTA, and microperimetry will be repeated once more after 4 months from the vitrectomy.
  Arms: Silicone oil group
Procedure: Pars plana vitrectomy with SF6 — Sulfur hexafluoride (SF6) will be used at the end of primary vitrectomy. OCT, OCTA, and microperimetry will be done 2 months and 4 months after surgery.
  Arms: Sulfur hexafluoride (SF6) group

SUMMARY:
Rhegmatogenous retinal detachment (RRD) is the separation of the neurosensory retina from the retinal pigment epithelium caused by the presence of a break that leads to the passage of fluid from the vitreous cavity into the potential subretinal space. It is a sight threatening disease, affecting largely people 50 years or older, with an annual incidence varying between 6.3 and 17.9 people per 100,000 population, and is unfortunately increasing. Although other surgical options do exist for the repair of primary RRD, pars plana vitrectomy (PPV) has clear advantages and is certainly effective in the treatment of these patients.

Several agents are used for intraocular tamponade following PPV for RRD. These agents are either silicone oil (SO) or gases like air, perfluoropropane (C3F8), sulfur hexafluoride (SF6), or perfluoroethane (C2F6).

In addition to the complications uniquely peculiar to using SO, research has found out that a reduction in retinal sensitivity on microperimetry was greater in SO tamponade in comparison with gas, as well as poorer visual outcome, microvasculature damage and affection of retinal layers including ganglion cell complex (GCC) in the SO group.

Even though many studies were done to compare between SO and intraocular gas tamponades with respect to many aspects, only one study compared the effects SO had on macular vasculature and anatomy in comparison with air and no study at all to date has compared the SO to SF6 gas in terms of retinal vascular changes, correlating them to thinning of GCC and macular sensitivity, which is precisely the main aim of the current study.

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachment (RRD) is the separation of the neurosensory retina from the retinal pigment epithelium (RPE) caused by the presence of a break that leads to the passage of fluid from the vitreous cavity into the potential subretinal space. It is a sight threatening disease, affecting largely people 50 years or older, with an annual incidence varying between 6.3 and 17.9 people per 100,000 population, and is unfortunately increasing. Although other surgical options do exist for the repair of primary RRD, viz. scleral buckling and pneumatic retinopexy, primary pars plana vitrectomy (PPV) has clear advantages and is certainly effective in the treatment of these patients, with a primary success rate of 85%, making it the leading management modality.

Several agents are used for intraocular tamponade following PPV for RRD, in order to provide surface tension across the retinal breaks thus preventing the ingress once more of fluid into the subretinal space, giving time for the permanent seal provided by the retinopexy done whether photocoagulation or cryopexy. These agents are either silicone oil (SO) or gases like air, perfluoropropane (C3F8), sulfur hexafluoride (SF6), or perfluoroethane (C2F6).

In addition to the complications uniquely peculiar to using SO, research has found out that a reduction in retinal sensitivity on microperimetry was greater in SO tamponade in comparison with gas, as well as poorer visual outcome, microvasculature damage and affection of retinal layers including ganglion cell complex (GCC) in the former group leading to the so-called Silicone Oil-Related Visual Loss (SORVL).

Even though many studies were done to compare between SO and intraocular gas tamponades with respect to many aspects, only one study by Zhou et al in 2020 compared the effects SO endotamponade had on macular vasculature and anatomy in comparison with sterilized air tamponade and no study at all to date has compared the SO to SF6 gas in terms of retinal vascular changes, correlating them to thinning of GCC and macular sensitivity, which is precisely the main aim of the current study.

ELIGIBILITY:
Inclusion Criteria:

* Primary rhegmatogenous retinal detachment

Exclusion Criteria:

* Macula-on retinal detachment
* Change of decision of type of endotamponade used intraoperatively
* Giant retinal tear
* Proliferative vitreoretinopathy worse than grade B
* Recent lens surgery within the previous 3 months prior to presentation
* Prior vitreoretinal surgery
* Macular hole
* Signs of epiretinal membrane
* Diabetic retinopathy
* Macular degeneration or other macular disorders
* Inferior retinal breaks between 4 and 8 o'clock
* History of uveitis
* History of glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Macular perfusion - FAZ | At 2 and 4 months following primary vitrectomy
  Comparison of foveal avascular zone area between the different treatment arms as a measure of macular perfusion.
Macular perfusion - SVP | At 2 and 4 months following primary vitrectomy
  Comparison of superficial retinal capillary vascular density between the different treatment arms.
Macular perfusion - DVP | At 2 and 4 months following primary vitrectomy
  Comparison of deep retinal capillary vascular density between the different treatment arms.

SECONDARY OUTCOMES:
Macular sensitivity | At 2 and 4 months following primary vitrectomy
  Comparison of macular sensitivity between the different treatment arms using macular microperimetry.
Thickness of ganglion cell complex | At 2 and 4 months following primary vitrectomy
  Comparison of the thickness of ganglion cell complex in microns between the different treatment arms using optical coherence tomography (OCT)
Best corrected visual acuity | At 2 and 4 months following primary vitrectomy
  Comparison of best corrected visual acuity between the different treatment arms using standard Snellen charts.
Retinal reattachment rate | At 4 months following primary vitrectomy
  Comparison of single-operation anatomical success (retinal reattachment) rate between the different treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Mina S. Abdelmalak, MSc, Principal Investigator — Cairo University; Soheir M. Mahmoud, PhD, Study Chair — Cairo University; Ahmed A. Abdel Kader, PhD, Study Director — Cairo University; Asmaa M. Shuaib, PhD, Study Director — Cairo University; Ayman G. Elnahry, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Results will be posted on clinicaltrials.gov when the study is concluded.

REFERENCES:
- [Background] Hajari JN, Bjerrum SS, Christensen U, Kiilgaard JF, Bek T, la Cour M. A nationwide study on the incidence of rhegmatogenous retinal detachment in Denmark, with emphasis on the risk of the fellow eye. Retina. 2014 Aug;34(8):1658-65. doi: 10.1097/IAE.0000000000000104. PMID 24978666
- [Background] Mitry D, Charteris DG, Fleck BW, Campbell H, Singh J. The epidemiology of rhegmatogenous retinal detachment: geographical variation and clinical associations. Br J Ophthalmol. 2010 Jun;94(6):678-84. doi: 10.1136/bjo.2009.157727. Epub 2009 Jun 9. PMID 19515646
- [Background] Nielsen BR, Alberti M, Bjerrum SS, la Cour M. The incidence of rhegmatogenous retinal detachment is increasing. Acta Ophthalmol. 2020 Sep;98(6):603-606. doi: 10.1111/aos.14380. Epub 2020 Feb 21. PMID 32086859
- [Background] Barrie T. Debate overview. Repair of a primary rhegmatogenous retinal detachment. Br J Ophthalmol. 2003 Jun;87(6):790. doi: 10.1136/bjo.87.6.790. No abstract available. PMID 12770985
- [Background] Vaziri K, Schwartz SG, Kishor KS, Flynn HW Jr. Tamponade in the surgical management of retinal detachment. Clin Ophthalmol. 2016 Mar 16;10:471-6. doi: 10.2147/OPTH.S98529. eCollection 2016. PMID 27041988
- [Background] Scheerlinck LM, Schellekens PA, Liem AT, Steijns D, van Leeuwen R. Retinal sensitivity following intraocular silicone oil and gas tamponade for rhegmatogenous retinal detachment. Acta Ophthalmol. 2018 Sep;96(6):641-647. doi: 10.1111/aos.13685. Epub 2018 Mar 2. PMID 29498239
- [Background] Ma Y, Zhu XQ, Peng XY. Macular Perfusion Changes and Ganglion Cell Complex Loss in Patients with Silicone Oil-related Visual Loss. Biomed Environ Sci. 2020 Mar 20;33(3):151-157. doi: 10.3967/bes2020.021. PMID 32209173
- [Background] Zhou Y, Zhang S, Zhou H, Gao M, Liu H, Sun X. Comparison of fundus changes following silicone oil and sterilized air tamponade for macular-on retinal detachment patients. BMC Ophthalmol. 2020 Jun 22;20(1):249. doi: 10.1186/s12886-020-01523-9. PMID 32571251
- [Background] Christensen UC, la Cour M. Visual loss after use of intraocular silicone oil associated with thinning of inner retinal layers. Acta Ophthalmol. 2012 Dec;90(8):733-7. doi: 10.1111/j.1755-3768.2011.02248.x. Epub 2011 Sep 13. PMID 21914150
- [Background] Raczynska D, Mitrosz K, Raczynska K, Glasner L. The Influence of Silicone Oil on the Ganglion Cell Complex After Pars Plana Vitrectomy for Rhegmatogenous Retinal Detachment. Curr Pharm Des. 2018 Dec 8;24(29):3476-3493. doi: 10.2174/1381612824666180813115438. PMID 30101697
- [Background] Newsom RS, Johnston R, Sullivan PM, Aylward GB, Holder GE, Gregor ZJ. Sudden visual loss after removal of silicone oil. Retina. 2004 Dec;24(6):871-7. doi: 10.1097/00006982-200412000-00005. PMID 15579983
- [Background] Goker YS, Yuksel K, Turan MF, Sonmez K, Tekin K, Yilmazbas P. Segmental Analysis of Macular Layers in Patients With Rhegmatogenous Retinal Detachment Treated With Perfluoropropane or Silicon Oil. Ophthalmic Surg Lasers Imaging Retina. 2018 Jan 1;49(1):41-47. doi: 10.3928/23258160-20171215-06. PMID 29304265
- [Background] Moharram HM, Abdelhalim AS, Hamid MA, Abdelkader MF. Comparison Between Silicone Oil and Gas in Tamponading Giant Retinal Breaks. Clin Ophthalmol. 2020 Jan 15;14:127-132. doi: 10.2147/OPTH.S237783. eCollection 2020. PMID 32021077
- [Background] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387
- [Background] Abrams GW, Azen SP, McCuen BW 2nd, Flynn HW Jr, Lai MY, Ryan SJ. Vitrectomy with silicone oil or long-acting gas in eyes with severe proliferative vitreoretinopathy: results of additional and long-term follow-up. Silicone Study report 11. Arch Ophthalmol. 1997 Mar;115(3):335-44. doi: 10.1001/archopht.1997.01100150337005. PMID 9076205
- [Background] Krzystolik MG, D'Amico DJ. Complications of intraocular tamponade: silicone oil versus intraocular gas. Int Ophthalmol Clin. 2000 Winter;40(1):187-200. doi: 10.1097/00004397-200040010-00018. No abstract available. PMID 10713925